CLINICAL TRIAL: NCT01903018
Title: A Multicenter, Phase II/III Study to Assess Radiation Induced Mucositis in Subjects With Locally Advanced Squamous Cell Carcinoma of the Head and Neck Administered Cisplatin and Radiation With or Without P276-00
Brief Title: A Study to Assess Radiation Induced Mucositis in Patients of Head and Neck Cancer Administered Chemo-Radiation With or Without P276-00
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P276-00/64/11
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Radiation Induced Mucositis in Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — P276-00; Radiotherapy; Cisplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- P276-00 (Experimental)
  Interventions: Drug: P276-00; Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: P276-00
Radiation: Radiation Therapy
Drug: Cisplatin

SUMMARY:
A Clinical Study to Assess Radiation Induced Mucositis in Subjects with Locally Advanced Squamous Cell Carcinoma of the Head and Neck

DETAILED DESCRIPTION:
A Multicenter, Phase II/III Study to Assess Radiation Induced Mucositis in Subjects with Locally Advanced Squamous Cell Carcinoma of the Head and Neck Administered Cisplatin and Radiation with or without P276-00

The Phase II component will be a single arm, open label, multicenter study to assess RIM in subjects with locally advanced SCCHN treated with P276-00 in combination with radiation therapy and cisplatin. '

The Phase III component will be a randomized, assessor blinded, multicenter, two-arm study to compare the time to onset of WHO Grade ≥ 3 RIM in subjects with locally advanced SCCHN (OC, OP, HP, and L) who are receiving definitive CRT for treatment of their malignancy. Subjects receiving definitive CRT will receive weekly intravenous cisplatin administered during radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to give an informed consent for the study.
2. Pathologically (histologically or cytologically) confirmed (from primary tumor and/or lymph nodes), non-metastatic diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx eligible for treatment with concomitant chemoradiation as first-line treatment; subjects with a history of surgical management are not eligible
3. Have a plan to receive a continuous course of radiation (3DRT or IMRT) as single daily fractions of 2.0 Gy, with a cumulative radiation dose between 66 and 70 Gy. Planned radiation treatment fields must include at least 2 oral sites (maxillary or mandibular labial mucosa, right or left buccal mucosa, right or left floor of the mouth, ventral tongue, right or left lateral tongue, or soft palate), with each site receiving more than equal to 50 Gy
4. Have a plan to receive a standard cisplatin regimen administered weekly (30 to 40 mg/m2)
5. Have an Eastern Co-operative Oncology Group (ECOG) performance status less than equal to 2
6. Males or females aged 18 years or older
7. Pre-treatment dental procedures must be completed with recovery and the prophylactic insertion of gastric feeding tubes (if planned) prior to entry into the study
8. Adequate bone marrow function measured within two weeks prior to enrollment based upon CBC/differential, defined as follows:

   1. Absolute neutrophil count (ANC) more than equal to 1,500 cells/mm3
   2. Platelets more than equal to 100,000 cells/mm3
   3. Hemoglobin (Hb) more than equal to 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hb more than equal to 8.0 g/dl prior to the start of RT is acceptable)
9. Adequate hepatic function measured within two weeks prior to enrollment defined as follows

   1. Bilirubin less than equal to 1.5 mg/dl
   2. AST less than equal to 2 times ULN
   3. ALT less than equal to 2 times ULN
10. Adequate renal function measured within two weeks prior to enrollment and defined as follows

    1. Serum creatinine less than equal to 1.5 mg/dl
    2. Creatinine clearance (CC) more than equal to 60 ml/min determined by 24-hour urine collection or estimated by the Cockcroft-Gault formula:
11. Have a negative serum pregnancy test for women of childbearing potential at time of screening and negative urine pregnancy test within 72 hrs prior to first dose of study drug

Exclusion Criteria:

1. Tumor of the lips, sinuses, salivary glands, nasopharynx, or unknown primary tumor
2. Metastatic disease (M1) Stage IVC as per the AJCC, 7th edition
3. Prior radiation to the head and neck
4. Have undergone induction CT
5. History of malignant tumors other than HNC (except non-melanoma skin cancer) unless disease free for a minimum of 3 years
6. Severe co-morbidity, defined as:

   1. Symptomatic and/or uncontrolled cardiac disease, New York Heart Association Classification III or IV
   2. Acute myocardial infarction within the last 6 months
   3. Acute bacterial or fungal infection requiring systemic antibiotics at the time of enrollment
   4. Subjects known to be seropositive for human immunodeficiency virus (HIV) or subjects with Acquired Immune Deficiency Syndrome (AIDS), known current acute or chronic Hepatitis B, known Hepatitis C (antigen positive), or hepatic cirrhosis
   5. Subjects with active tuberculosis
   6. Collagen vascular disease, such as scleroderma, as this is thought to predispose subjects to increased risk for radiation-associated toxicities
7. Have used any other investigational drug therapy within 1 month prior to Day 1 of study drug administration or non-recovery (to Grade less than equal to 1) from adverse effects of the investigational agent received prior to this period
8. Prior allergic reaction to any of the agents administered during the course of treatment
9. Have QTcF more than equal to 450 msec at screening
10. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of severe Radiation Induced Mucositis (WHO grade >=3) | Week 15
  For Phase2, to assess the incidence of severe (WHO Grade >=3) Radiation Induced Mucositis (RIM)occurring up to a cumulative radiation dose of 66 Gray (Gy) based on the WHO mucositis scale in subjects with locally advanced squamous cell carcinoma of the head and neck (SCCHN) treated with cisplatin and radiotherapy plus P276-00
  * For Phase 3
  * To assess and compare the incidence of severe (WHO Grade>=3) Radiation Induced Mucositis (RIM) occurring up to a cumulative radiation dose of 54 Gy based on the WHO mucositis scale
  * To assess and compare the incidence of severe (WHO Grade>=3) RIM occurring up to a cumulative radiation dose of 66 Gy based on the WHO mucositis scale in subjects with locally advanced SCCHN treated with cisplatin and radiotherapy plus P276-00 or cisplatin and radiotherapy (the two treatment arms).

SECONDARY OUTCOMES:
Time to onset of severe RIM (WHO Grade ≥ 3) | Week 15
  To evaluate the time to onset of severe RIM (WHO Grade>=3) as defined by the number of days between start of study treatment and the first time that WHO Grade 3 or 4 mucositis was observed (regardless of whether it had been Grade 0,1 or 2 previously)
Duration of severe RIM (WHO Grade>=3) | Week 15
  To assess the duration of severe RIM (WHO Grade>=3) as defined by the number of days from the onset of severe RIM as defined above, to the day when severe RIM resolved (first time when WHO Grade 0, 1, or 2 was observed)
Progression-Free Survival (PFS) | 1year
  To assess Progression-Free Survival (PFS)
Overall Survival (OS) | 1year
  To assess Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Sarbani Ghosh Laskar, MD, Principal Investigator
Locations (7):
- India (7):
  - Bharat Cancer Hospital & Research Institute, Surat, Gujarat
  - Sri Venkateshwara Hospitals, Bangalore, Karnataka
  - Mazumdar Shaw Cancer Center, Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Curie Manavta Cancer Centre, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Meenakshi Mission Hosp. & Res. Centre, Madurai, Tamil Nadu